CLINICAL TRIAL: NCT03635658
Title: Assessment of Guided Bone Regeneration in Augmentation of Horizontally Atrophic Maxillary Ridge Using Collagen Membrane Versus Using Titanium Mesh: a Randomized Controlled Clinical Trial
Brief Title: Assessment of GBR in Augmentation of Horizontally Atrophic Maxillary Ridge Using Collagen Membrane Versus Using Titanium Mesh
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Randa khaled Ismail, assistant lecturer in oral and maxillofacial department cairo university, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEBD-CU-2018-08-12
Record Dates: First submitted 2018-08-13; First posted 2018-08-17 (Actual); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Horizontal Ridge Deficiency

STUDY DESIGN:
Intervention Model Description: the participants are divided into two groups one control and the other is the intervention
Masking Description: because the two interventions used in this trial are clearly different and easily recognized by the investigator and the participants. neither the participant nor the investigator could be blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- titanium mesh (Active Comparator): using non resorbable titanium mesh to fix and cover the onlay bone graft mixture to the atrophic maxillary ridge.
  Interventions: Procedure: titanium mesh
- collagen membrane(Sausage technique) (Experimental): using resorbable collagen membrane with the sausage technique to fix the onlay bone graft mixture to the resorbed atrophic maxillary ridge
  Interventions: Procedure: collagen membrane (Sausage technique)

INTERVENTIONS:
Procedure: titanium mesh — the non resorbable titanium mesh is used to fix the 1:1 mixture of autograft and xenograft particulate bone on the severely atrophies maxillary ridge.
  Arms: titanium mesh
Procedure: collagen membrane (Sausage technique) — the resorbable collagen membrane is used to fix the 1:1 mixture of autograft and xenograft particulate bone on the severely atrophies maxillary ridge.
  Arms: collagen membrane(Sausage technique)

SUMMARY:
this study is aiming to Assess postoperative complications and bone quality and quantity in augmentation of horizontally atrophic maxillary ridge using a 1:1 mixture of autograft and xenograft particulate bone covered with collagen membrane with the new Sausage technique™ versus using the same mixture covered with titanium mesh.

DETAILED DESCRIPTION:
patients with atrophic maxillary ridge < 4 mm will be selected in this study for augmentation for future implant placement. The full thickness flap will be elevated including one extra tooth on each side of the edentulous area or if completely edentulous 5 mm on each side.. the bone bed will be prepared by cleaning any debris and Multiple decortication holes will be performed with a 2.0 mm round bur. the harvested bone from the chin is then mixed with the xenograft with ratio 1:1 and then put on the recipient site and will be covered with a collagen membrane with the Sausage technique (intervention group) and the other group the graft will be covered with titanium mesh (control group).

flap is repositioned and sutured. followup for 6 months and then CBCT is done. Reopening after 6 months, core biopsy is taken by a 2 mm thickness trephine from the healed augmented bone at the site of implant placement and will be sent for histomorphometric analysis and the bone thickness (buccolingual ) dimension is measured using a caliper and from the CBCT (cone beam CT) the bone width gain will be calculates and recorded.

postoperative complications( infection, wound dehiscence or membrane exposure) will be monitored and recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with horizontal atrophied maxillary ridge (thin ridge) less than 4mm.
2. All ages and both sexes were included in this study.
3. Patients should be free from any systemic disease that may affect normal healing of bone, and predictable outcome.
4. Patients with physical and psychological tolerance

Exclusion Criteria:

1. Patients with high risk systemic diseases like uncontrolled diabetes mellitus. As uncontrolled diabetes mellitus has a negative impact on normal bone healing. 8
2. Heavy smokers.4
3. Alcohol or drug abuse
4. Gingival bleeding or full mouth plaque index ≥ 25%.4
5. Patients with physical and psychological intolerance. As psychological stress will affect the immune system and patient's fitness including healing capacity. 9
6. Unavailability for regular follow-ups

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-10-01 (Estimated); Primary Completion 2019-03-01 (Estimated); Study Completion 2020-10-01 (Estimated)

PRIMARY OUTCOMES:
membrane exposure | within 3 weeks
  clinical postoperative complications as flap dehiscence and membrane exposure into the oral cavity, its a binary outcome (yes/No) examined and recorded by the investigator.
infection | 10 days
  suppuration collection related to the membrane and flap, its a binary outcome (yes/No) examined and recorded by the investigator.
inflammation | 10 days
  redness and tenderness of the flap, its a binary outcome (yes/No) examined and recorded by the investigator.

SECONDARY OUTCOMES:
bone width gain | at 6 months
  the amount of bone gained( in millimeter) after augmentation compared to the initial ridge thickness measured clinically using a caliper 2 mm below the crest of the ridge, and radiographically using the Planmeca Promax 3D CBCT unit which will be viewed on planmeca romexis software to calculate the measures needed in millimeter by the outcome assessor.
bone quality | at 6 months
  histomorphometric analysis of the bone biopsy taken from the augmented bone to show the quality of the formed bone and the percentage of every type of tissue formed in the specimen taken( unit is area percentage %)